CLINICAL TRIAL: NCT05787392
Title: Chamas For Change: A Gender-Responsive And Microfinance-Based Approach To Empowering Women And Building Resilience To Health Emergencies in Kenya
Brief Title: Chamas for Change: Impact of the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Moi University (Other)
Collaborators: International Development Research Centre, Canada (Other Government); University of British Columbia (Other); Indiana University (Other); University of Toronto (Other)
Responsible Party: Principal Investigator, Astrid Christoffersen-Deb, Assistant Professor, Moi University
Other Study IDs: MoiU7
Record Dates: First submitted 2023-03-23; First posted 2023-03-28 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Gender Equity
Keywords: participatory research; Gender equity; maternal and child well-being; Kenya; Mixed-methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Completed Chamas program: women who participated in Chamas throughout the pandemic
  Interventions: Behavioral: Chamas cha MamaToto program
- Did not complete Chamas program: women who left Chamas during the pandemic
  Interventions: Behavioral: Chamas cha MamaToto program
- Did not participate in Chamas program: women whose communities were randomized to not receive the Chamas intervention

INTERVENTIONS:
Behavioral: Chamas cha MamaToto program — Chamas is a community health volunteer (CHV)-led group programme that engages women during pregnancy and the first 1000 days of their child's life. The strategy focuses on promoting maternal, newborn, and child health (MNCH) by providing health education, peer support, and opportunities to access financial capital, all while addressing inequities that perpetuate poor outcomes.
  Groups: Completed Chamas program; Did not complete Chamas program

SUMMARY:
In Kenya, the chamas strategy (a peer support approach aimed at improving MNCH and reducing gender and social inequalities) has been shown to significantly improve maternal and child health outcomes while also providing social and financial support to participating women. However, the COVID-19 pandemic caused significant disruptions in women's work and MNCH services around the world due to reallocation of health care resources, COVID-19 fears, transportation restrictions, and lockdowns. These consequences appeared to disproportionately affect the poor, particularly poor women. The purpose of this participatory action design study is to determine how Chamas participation intersected with other factors to mitigate the effects of the COVID-19 pandemic on the health and economic well-being of women and children.

DETAILED DESCRIPTION:
The study objectives are:

To evaluate the effect of Chama participation on mitigating the effects of the pandemic on social and gender equity.

* Impact on economic status (assessed using the changes in the Poverty Probability index scores)
* Impact on health service utilization and behaviours (assessed using enrollment in the national health insurance scheme, number of ANC visits attended, facility delivery, maternal death, newborn death, infant death, exclusive breastfeeding, number of children fully immunized at age 1)
* Social attitudes and well-being (assessed using, attitude towards harsh punishment of children, level of parental stress)
* COVID-19 related information (assessed using COVID-19 infection, COVID-19 vaccination, and effects of COVID restrictions)

To use an equity-centered design process and narrative approach to share research findings.

The research team intends to evaluate women's experiences during the pandemic using a mixed method approach and a participatory action design method. The focus will be on 3 study cohorts: (1) women who participated in Chamas throughout the pandemic, (2) women who left Chamas during the pandemic, (3) women whose communities were randomized to not receive the Chamas intervention. To better understand the effects of Chama participation on study outcomes, we will conduct an interviewer-administered survey among the described cohorts of women. This will be followed by qualitative studies to contextualize the study findings and investigate gender dynamics as social processes. Focus group discussions (FGDs) and key informant interviews (KIIs) will be conducted to further investigate our study cohort's experiences during the pandemic and identify strategies used by participants to mitigate the negative effects of the pandemic and its associated restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Women who participated in the 2021 Chamas study in Western Kenya

Exclusion Criteria:

* Women who did not participate in the 2021 study.

Ages: 15 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes
Study Population: This research will be conducted in Trans-Nzoia County among the 1400 women that participated in the 2021 RCT study. The following groups will be included in our study population.
  * RCT women who participated in Chamas throughout the pandemic.
  * Women who left Chamas after March 12, 2020, the date the first case of COVID-19 was discovered in Kenya.
  * Women whose communities were randomly assigned not to use Chamas during the RCT.
  * CHVs in communities that had or did not have Chamas operating during the pandemic.
  * County health officials.
  * Fathers participating in Chama cha Babatoto.
  * Adolescent girls are currently participating in Chamas adapted for adolescents.
Sampling Method: Non-Probability Sample
Enrollment: 444 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-03-13 (Estimated); Study Completion 2025-03-13 (Estimated)

PRIMARY OUTCOMES:
Economic Status | 1 year
  Impact of COVID-19 pandemic on the women's economic well-being based on Poverty property Index (PPI) scores obtained from 10 questions in the questionnaire. The PPI is a relative scale in which each response is assigned a value, and the sum of the values is the participant's PPI score. The participant's PPI is then compared with the country level score using the "look-up table" for the country (Kenya) to determine the participant's likelihood of being poor. The investigators will compare the PPI scores at the post-pandemic period between the three cohorts in the study.

SECONDARY OUTCOMES:
Health insurance uptake | 1 year
  Enrolment in health insurance based on questionnaire response.
Health service utilization | 1 year
  Use of health services during the COVID-19 pandemic based on questionnaire response to questions assessing use of healthcare services during the COVID-19 pandemic.
Social impact of COVID19 | 1 year
  Parenting stress based on parental stress index scale scores in questionnaire. Overall possible scores on the scale range from 18 - 90. The higher the score, the higher the measured level of Parental stress
Attitudes towards Harsh punishment | 1 year
  Attitude to child punishment based on questionnaire response.
COVID-19 experiences of key informants | 1 year
  Experiences of the community during the COVID pandemic from the perspective of key informants will be explored based on qualitative interviews. Questions to explore how different genders experienced the pandemic will be specifically explored. The gender considerations will include an assessment of how gender interacts with resource access, the roles each gender plays in society, societal expectations, and power dynamics. It also includes evaluating the ways in which gender power relations manifest to create inequities and/or differences in experiences during the pandemic.
COVID-19 experiences | 1 year
  Experiences of the community during the COVID pandemic from the perspective of the three cohorts of women in the study will be explored based on qualitative focus group discussions. Questions to explore how different genders experienced the pandemic will be specifically explored. The gender considerations will include an assessment of how gender interacts with resource access, the roles each gender plays in society, societal expectations, and power dynamics. It also includes evaluating the ways in which gender power relations manifest to create inequities and/or differences in experiences during the pandemic.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Songok, Principal Investigator — AMPATH Kenya; Sammy Masibo, Study Director — Trans Nzoia county government; Michael Scanlon, Study Director — Indiana University; Laura Ruhl, Study Director — Indiana University; Julie Thorne, Study Director — University of Toronto; Violet Naanyu, Study Director — Moi University
Locations (2):
- Kenya (2):
  - Trans Nzoia county, Kiminini
  - Trans-Nzoia County, Kitale

DOCUMENTS (1):
  • Study Protocol (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT05787392/Prot_001.pdf